CLINICAL TRIAL: NCT05249244
Title: A Real World Study of the Treatment of Locally-inoperable Advanced or Advanced Metastatic Gastric Adenocarcinoma With Huachansu
Brief Title: A Real World Study of the Treatment of Gastric Adenocarcinoma With Huachansu
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: China Resources Sanjiu Medical & Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ICM-HCS-CR01
Record Dates: First submitted 2022-01-20; First posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Gastric Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- observation group: huachansu oral preparation (tablet, capsule) was used.
- control group: huachansu was not used.

SUMMARY:
To evaluate the efficacy and safety of huachansu oral preparation in the treatment of inoperable locally advanced or advanced metastatic gastric adenocarcinoma, including gastric esophageal adenocarcinoma.

DETAILED DESCRIPTION:
In this multicenter, controlled, retrospective, real-world study, the original medical records of participants diagnosed with inoperable locally advanced or advanced metastatic gastric adenocarcinoma (including gastric esophageal junction adenocarcinoma) receive treatment in research centers from January 1, 2014 to December 31, 2019 were collected. To evaluate the efficacy and safety of oral huachansu in the systematic treatment of locally advanced or advanced metastatic gastric adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

Only patients who meet all the following criteria are included in the study:

1. Diagnosed with gastric adenocarcinoma (including gastric esophageal junction adenocarcinoma) by histopathology or cytology at the enrolled centers From January 1, 2014 to December 31, 2019.
2. Stage of disease (clinical or pathological stage) is locally advanced or advanced (stage IIIB-IV) .
3. The doctor judged that the tumor tissue was unresectable.
4. At least two medical records.
5. At least one huachansu oral preparation (tablet, capsule) was used during treatment (observation group only) .

Exclusion Criteria:

Patients who meet any of the following criteria are not allowed to enter the test:

1. Lack of clinical data related to important research indicators (survival).
2. Refusal to cooperate with follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with locally inoperable advanced or advanced metastatic gastric adenocarcinoma (including gastric esophageal junction adenocarcinoma) admitted to the study centers between January 1, 2014 and December 31, 2019.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
OS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  overall survival
AE;SAE | 1 year, year 1
  adverse event;Serious Adverse Event

SECONDARY OUTCOMES:
ADR;SADR | 1 year, year 1
  Adverse Drug Reaction;Serious Adverse Drug Reaction

OTHER OUTCOMES:
ORR | through study completion
  ORR=CR+PR
DCR | through study completion
  DCR=CR+PR+SD
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  progression-free survival
BMI | through study completion
  BMI=weight（kg）/height²（m²）
Use of painkillers during treatment | through study completion
  Proportion of patients using painkillers during treatment

CONTACTS AND LOCATIONS:
Overall Officials: kangsheng gu, Principal Investigator — The First Affiliated Hospital of Anhui Medical University
Locations (1):
- The First Affiliated Hospital of Anhui Medical University, Hefei, China

IPD SHARING:
Plan to Share IPD: No